CLINICAL TRIAL: NCT01172353
Title: Hydration With Sodium Bicarbonate for Prevention of Contrast-Induced Nephropathy: A Multicenter Clinical Trial
Brief Title: Sodium Bicarbonate for Prevention of Contrast-Induced Nephropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Sao Lucas da PUCRS (Other)
Responsible Party: Principal Investigator, Vitor Osorio Gomes, MD, PhD, Hospital Sao Lucas da PUCRS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSaoLucas
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Results first posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-01

CONDITIONS: Renal Failure
Keywords: contras-induced nephropathy
MeSH Terms: conditions — Renal Insufficiency | interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- sodium bicarbonate (Experimental): hydration with sodium bicarbonate
  Interventions: Drug: sodium bicarbonate
- saline (Active Comparator): hydration with saline 1ml/Kg/h for 6 hours
  Interventions: Drug: saline

INTERVENTIONS:
Drug: sodium bicarbonate — hydration with sodium bicarbonate 1ml/Kg/h for 6 hours
  Arms: sodium bicarbonate
Drug: saline — hydration with saline 1ml/Kg/h for 6 hours
  Arms: saline

SUMMARY:
The purpose of this study is to determine whether hydration with sodium bicarbonate is superior to hydration with saline to prevent contrast-induced nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* serum creatinine > 1.1 mg/dL
* glomerular filtration rate (GFR) < 50 mL/min

Exclusion Criteria:

* age < 18 years
* use of radiographic contrast media during the last 21 days
* history of dialysis
* cardiac insufficiency class III-IV
* emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2004-07; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- São Lucas Hospital - PUCRS University, Porto Alegre, Rio Grande do Sul, Brazil

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sodium Bicarbonate | Saline
Started | 150 | 151
Completed | 150 | 151
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Bicarbonate | Saline | Total
Number analyzed (Participants) | 150 | 151 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (12) | 64.5 (12) | 64.3 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 38 | 84
  Male | 104 | 113 | 217
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 140 | 140 | 280
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 150 | 151 | 301

OUTCOME MEASURES:

1. Primary Outcome: Contrast-induced Nephropathy
Description: rise in serum creatinine >0,5mg/dl
Time Frame: 48 hours
Measure: Number; unit: percentage of contrast nephropaty
Arm/Group | Sodium Bicarbonate | Saline
Number analyzed (Participants) | 150 | 151
percentage of contrast nephropaty | 6.1 | 6.0

2. Secondary Outcome: Dialysis During Hospitalization
Time Frame: During hospitalization
Measure: Number; unit: participants
Arm/Group | Sodium Bicarbonate | Saline
Number analyzed (Participants) | 150 | 151
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Sodium Bicarbonate | Saline
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/151
Other Adverse Events (participants affected / at risk) | 0/150 | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No